CLINICAL TRIAL: NCT00001797
Title: Randomized Double-Blind Placebo-Controlled Trial Using Recombinant Human Interleukin-10 for Moderate-to-Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 990027; 99-C-0027
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-12

CONDITIONS: Psoriasis
Keywords: Cytokines; Immunomodulation; Inflammation; Skin; Therapy
MeSH Terms: conditions — Psoriasis; Inflammation

INTERVENTIONS:
Drug: Recombinant human interleukin-10

SUMMARY:
Several studies have documented an essential role for interleukin-10 (IL-10) in preventing prolonged and exaggerated immune responses to antigens and irritants. Psoriasis, a relatively common disease, is characterized by T cell-mediated inflammation in affected skin. In this study, the safety, tolerance, immunologic effects, and clinical activity of subcutaneous (SC) recombinant human (rh) IL-10 will be evaluated in patients with moderate-to-severe psoriasis. There will be 2 groups of patients, randomized to receive either 20 ug/kg rhIL-10 SC 3 times weekly (20 patients) or SC placebo (10 patients). This double-blind phase will continue for a total of 12 weeks and the principal evaluation will be the comparison between baseline and 12 week Psoriasis Area Severity Index (PASI) scores. Patients will come for an initial screening visit at day 0, and at weeks 1, 2, 4, 6, 8, and 12, with follow-up visits at weeks 16 and 20.

All patients will be offered rhIL-10 at 12 weeks (following the blinded portion of the study protocol). Patients initially receiving active medication who wish to continue rhIL-10 therapy will be kept on the drug. This open-label portion of the study will continue for an additional 12 weeks. Patients continuing with active drug will be evaluated at weeks 14, 16, 20, and 24.

Skin disease activity and toxicity will be assessed and recorded throughout the study. In addition, research studies will include functional assays to assess cytokine secretion and immunologic function of peripheral blood cells and immunohistochemical characterization of the inflammatory cells in skin.

DETAILED DESCRIPTION:
Several studies have documented an essential role for interleukin-10 (IL-10) in preventing prolonged and exaggerated immune responses to antigens and irritants. Psoriasis, a relatively common disease, is characterized by T cell-mediated inflammation in affected skin. In this study, the safety, tolerance, immunologic effects, and clinical activity of subcutaneous (SC) recombinant human (rh) IL-10 will be evaluated in patients with moderate-to-severe psoriasis. There will be 2 groups of patients, randomized to receive either 20 (micro)g/kg rhIL-10 SC 3 times weekly (20 patients) or SC placebo (10 patients). This double-blind phase will continue for a total of 12 weeks and the principal evaluation will be the comparison between baseline and 12 week Psoriasis Area Severity Index (PASI) scores. Patients will come for an initial screening visit at day 0, and at weeks 1, 2, 4, 6, 8, and 12, with follow-up visits at weeks 16 and 20.

All patients will be offered rhIL-10 at 12 weeks (following the blinded portion of the study protocol). Patients initially receiving active medication who wish to continue rhIL-10 therapy will be kept on the drug. This open-label portion of the study will continue for up to an additional 12 weeks. Patients continuing with active drug will be evaluated at weeks 14, 16, 20, and 24.

Skin disease activity and toxicity will be assessed and recorded throughout the study. In addition, research studies will include functional assays to assess cytokine secretion and immunologic function of peripheral blood cells and immunohistochemical characterization of the inflammatory cells in skin.

ELIGIBILITY:
Able to provide informed consent to all aspects of the study after full information is provided.

Age equal to or between 18 and 65 years.

Moderate-to-severe stable plaque psoriasis of at least 6 months duration as defined by the following criteria: 1) Classic psoriatic skin lesions with or without nail involvement, 2) Psoriasis Area and Severity Index score greater than 10(i), 3) Total body surface area involved greater than 10%.

Weight less than 242 pounds.

Must be able to self-administer medication (subcutaneous injection) or arrange for administration.

No unstable psoriatic disease, including erythrodermic, pustular, and palmar/plantar variants.

No use of topical medications for psoriasis (except for bland emollients) during 2 weeks prior to study entry.

No use of systemic medications for psoriasis during 1 month prior to study entry.

No patients with an ECOG or Zubrod Performance Status Scale greater than 2.

No patients with acute or chronic infections requiring antimicrobial therapy or serious viral (e.g., hepatitis, herpes zoster, or HIV) or fungal infections as the effects of IL-10 on the immune system not completely elucidated and treatment could pose additional risk to the patient. Patients with a positive PPD who have not received antituberculous therapy may be excluded, if in the opinion of an infectious consultant, IL-10 treatment is contraindicated.

No patients receiving disease modifying anti-inflammatory drugs (methotrexate, sulfasalazine, gold, hydroxychloroquine, cyclosporin, azathioprine, cyclophosphamide, chlorambucil, retinoids, vitamin D). Such drugs will be discontinued at least 4 weeks prior to randomization.

No pregnant females, nursing mothers, or patients of childbearing age not practicing birth control, since the risks to the unborn fetus and newborn child are unknown.

No previous history of malignancy or current malignancy other than satisfactorily treated basal-squamous cell carcinoma or in situ cervical carcinoma.

No confounding medical illness that in the judgment of the investigators would pose added risk for study participants (e.g., hepatic, hematologic [e.g., hematocrit less than or equal to 28% or platelet counts less than 100,000/ml], neurologic, renal, or pulmonary disease).

No patients with serum creatinine greater than 1.8 or creatinine clearance (CrCl) less than 50 ml/min.

No patients with abnormal liver function tests (e.g., serum glumatic oxalacetic transaminase, serum glutamic pyruvic transaminase or alkaline phosphatase levels greater than 2.5x upper limit of normal (UNL) and/or bilirubin levels 1.5x UNL).

No current alcohol or drug abuse.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Start 1999-01; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Uyemura K, Yamamura M, Fivenson DF, Modlin RL, Nickoloff BJ. The cytokine network in lesional and lesion-free psoriatic skin is characterized by a T-helper type 1 cell-mediated response. J Invest Dermatol. 1993 Nov;101(5):701-5. doi: 10.1111/1523-1747.ep12371679. PMID 7693825
- [Background] Schlaak JF, Buslau M, Jochum W, Hermann E, Girndt M, Gallati H, Meyer zum Buschenfelde KH, Fleischer B. T cells involved in psoriasis vulgaris belong to the Th1 subset. J Invest Dermatol. 1994 Feb;102(2):145-9. doi: 10.1111/1523-1747.ep12371752. PMID 8106745
- [Background] Nestle FO, Turka LA, Nickoloff BJ. Characterization of dermal dendritic cells in psoriasis. Autostimulation of T lymphocytes and induction of Th1 type cytokines. J Clin Invest. 1994 Jul;94(1):202-9. doi: 10.1172/JCI117308. PMID 8040262